CLINICAL TRIAL: NCT00104130
Title: A Phase 2 Study of KOS-862 Administered Intravenously Weekly for 3 Weeks Every 4 Weeks, in Patients With Hormone Resistant Prostate Cancer Who Have Progressed Following Initial Therapy for Metastatic Disease
Brief Title: Study of KOS-862 (Epothilone D) in Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOS-202/NO18401
Record Dates: First submitted 2005-02-23; First posted 2005-02-24 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-09

CONDITIONS: Prostate Cancer
Keywords: prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — desoxyepothilone B

INTERVENTIONS:
Drug: KOS-862

SUMMARY:
The purpose of this trial is to study KOS-862 in men with metastatic prostate cancer who have failed a docetaxel-containing regimen.

DETAILED DESCRIPTION:
This study is a Phase 2, single arm study of KOS-862 in men with metastatic prostate cancer who have failed a docetaxel-containing regimen. PSA response is the primary end-point and objective responses will be checked as available.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Metastatic disease.
* One previous treatment including docetaxel (Taxotere).
* At least 3 weeks since last surgery/radiation/chemotherapy
* ECOG Performance Status of 0, 1 or 2

Exclusion Criteria:

* Active brain metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53
Dates: Start 2004-12; Study Completion 2005-02

PRIMARY OUTCOMES:
prostate cancer
prostate-specific antigen (PSA) response

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Kaiser Permanente Medical Center, Vallejo, California
  - Georgia Cancer Specialists, Tucker, Georgia
  - University of Maryland Medical System, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Kaiser Permanente NW Oncology Clinic, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington